CLINICAL TRIAL: NCT05081518
Title: Interventional, Randomized, Double-blind, Crossover, Placebo-controlled, Multiple-dose Lu AG06466 Phase 1 B Study in Patients With Focal Epilepsy Using EEG and PSG to Investigate Its Pharmacodynamic Effects on Prolonged Period of Inter- Icterical Spikes, Sleep and Neuroinflammation
Brief Title: A Study of Lu AG06466 in Participants With Treatment Resistant Focal Epilepsy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to enrolment challenges
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19367A
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Lu AG06466-Placebo (Experimental): Participants will receive Lu AG06466 capsules once daily (QD) at a low dose for 4 days (Days 1 to 4), medium dose for 4 days (Days 5 to 8), and high dose for 21 days (Days 9 to 29) in treatment period 1. Participants will receive matching placebo capsules from Day 1 to Day 29 in treatment period 2. Each treatment period will be separated by a washout period of 7 to 11 days.
  Interventions: Drug: Lu AG06466; Drug: Placebo
- Sequence 2: Placebo-Lu AG06466 (Experimental): Participants will receive matching placebo capsules QD from Day 1 to Day 29 in treatment period 1. Participants will receive Lu AG06466 capsules QD at a low dose for 4 days (Days 1 to 4), medium dose for 4 days (Days 5 to 8), and high dose for 21 days (Days 9 to 29) in treatment period 2. Each treatment period will be separated by a washout period of 7 to 11 days.
  Interventions: Drug: Lu AG06466; Drug: Placebo

INTERVENTIONS:
Drug: Lu AG06466 — Lu AG06466 - capsule
Drug: Placebo — Placebo - capsule

SUMMARY:
The main purpose of this study is to investigate effects of Lu AG06466 on seizure activity after increasing daily doses during 4 weeks in participants with an implanted responsive neurostimulation system.

DETAILED DESCRIPTION:
This crossover study consists of 2 treatment periods, each of 29 days duration. On Day -1 of treatment period 1, eligible participants will be randomized (1:1) to a sequence of treatments (either Lu AG06466-placebo or placebo-Lu AG06466).

ELIGIBILITY:
Key Inclusion Criteria:

* The participant must have had the responsive neurostimulation system (RNS®) System implanted for more than 1 year and medically intractable focal onset epileptic seizures (history of persistent seizures refractory to 2 or more anti-epileptic drugs [AEDs]), with seizures from all foci represented in the implanted RNS electrodes.
* The participant is required to have a continuous period of at least 2 months prior to the Screening Visit with constant RNS stimulation settings as well as stable AED (that is, 60 days with no dose adjustments of more than 25%) as determined by medical history and the Patient Data Management System (PDMS). There must be at least 24 recorded long episodes available for review since last change of RNS detection setting.
* The participant is required to have approximately 7 or more long episodes per week, as assessed as an average over the last 2 months prior to the Screening Visit.
* The participant is required to have a demonstrated history of compliance with RNS scanning and uploading procedure in the past year (less than 20% missing long episode counts on the PDMS).

Key Exclusion Criteria:

* The participant has the RNS System implanted in other regions than the epileptic foci such as the thalamus.
* The participant has a RNS System with anticipated generator change in the coming 6 months.
* The participant has a cyclic pattern of long episodes in the last 2 months prior to the Screening Visit which exhibits, in the opinion of the investigator: a period of more than 3 weeks; and peak-to-trough differences of long episodes of more than half the peak level.
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological (apart from epileptic diagnosis), or psychiatric disease or other major disorder, which in opinion of the investigator may influence efficacy or safety aspects in the study.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Number of "Long Episodes" (Electrocorticographic [ECoG] Seizures) | Baseline (Day -1) up to Day 29 of each treatment period
  "Long Episodes" are abnormal events detected by the neurostimulator that do not return to baseline ECoG activity within a predefined period of time, typically 30 to 60 seconds. These often correspond to ECoG seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States